CLINICAL TRIAL: NCT04840459
Title: Use of Monoclonal Antibodies (Bamlanivimab and Casirivimab + Imdevimab) for the Treatment of Mild to Moderate COVID-19 in Non-Hospitalized Setting
Brief Title: Use of Monoclonal Antibodies for the Treatment of Mild to Moderate COVID-19 in Non-Hospitalized Setting
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohail Rao (Other)
Responsible Party: Sponsor-Investigator, Sohail Rao, President and CEO, DHR Health Institute for Research and Development
Organization: DHR Health Institute for Research and Development (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1686206
Record Dates: First submitted 2021-04-05; First posted 2021-04-12 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — bamlanivimab; casirivimab; imdevimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BAMLANIVIMAB (Experimental): The dosage of bamlanivimab in adults and pediatric patients 12 years of age and older weighing at least 40 kg is a single IV infusion of 700 mg bamlanivimab administered over at least 60 minutes
  Interventions: Biological: BAMLANIVIMAB
- CASIRIVIMAB + IMDEVIMAB (Experimental): 10 mL of casirivimab and 10 mL of imdevimab from each respective vial using two separate syringes and dilute together in the infusion bag containing 0.9% Sodium Chloride Injection
  Interventions: Biological: CASIRIVIMAB; Biological: IMDEVIMAB

INTERVENTIONS:
Biological: BAMLANIVIMAB — n. Bamlanivimab is a recombinant neutralizing human mIgG1? monoclonal antibody (mAb) to the spike protein of SARS-CoV-2, and is unmodified in the Fc region.
  Arms: BAMLANIVIMAB
Biological: CASIRIVIMAB — CASIRIVIMAB is a recombinant human mAbs which are unmodified in the Fc regions.
  Arms: CASIRIVIMAB + IMDEVIMAB
Biological: IMDEVIMAB — IMDEVIMAB is a recombinant human mAbs which are unmodified in the Fc regions.
  Arms: CASIRIVIMAB + IMDEVIMAB

SUMMARY:
No therapeutic agent is currently approved for the treatment of SARSCoV-2 infection. More importantly, no intervention is currently available to mitigate the progression of disease from mid/moderate to serve particularly in high risk patients. Recognizing this limitation and urgency of finding a treatment for COVID-19, the U.S. Food and Drug Administration (FDA) has issued an Emergency Use Authorization (EUA) to permit the emergencyuse of the unapproved product bamlanivimab or casirivimab + imdevimab for the treatment of mild to moderate coronavirus disease 2019 (COVID19) in adults and pediatric patients with positive results of direct SARS-CoV-2 viral testing who are 12 years of age and older weighing at least 40 kg, and who are at high risk for progressing to severe COVID-19 and/or hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. adults and pediatric patients with positive results of direct SARS-CoV-2 viral testing
2. 12 years of age and older weighing at least 40 kg
3. are at ":high risk" for progressing to severe COVID-19 and/or hospitalization

High risk is defined as patients who meet at least one of the following criteria:

1. Have a body mass index (BMI) >35
2. Have chronic kidney disease
3. Have diabetes
4. Have immunosuppressive disease
5. Are currently receiving immunosuppressive treatment
6. Are over 65 years of age
7. Are over 55 years of age AND have: cardiovascular disease, OR hypertension, OR chronic obstructive pulmonary disease/other chronic respiratory disease
8. Are 12 - 17 years of age AND have
9. BMI >85th percentile for their age and gender based on CDC o growth charts, ii. sickle cell disease OR iii. congenital or acquired heart disease OR iv. neurodevelopmental disorders, for example, cerebral palsy, OR a medical-related technological dependence, for example, tracheostomy, gastrostomy, or positive pressure ventilation (not related to COVID-19), OR

v. asthma, reactive airway or other chronic respiratory disease o that requires daily medication for control.

Exclusion Criteria

1. Younger than 12 years of age
2. Do not meet criteria to be classified as "high risk'

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Minimize and/or eliminate the number of patients with mild to moderate COVID-19 who are at high risk for progressing to severe COVID-19 and/or hospitalization. | two weeks
  Will record the number of participants who are prevented from progressing to sever infection.

OTHER OUTCOMES:
Determine Rate of Recovery after monoclonal antibody therapy | six weeks from monoclonal administration
  Participants will complete a questionnaire that will ask them to answer when symptoms started and how long after monoclonal antibody therapy did participants begin to feel better
Determine if if Hospitalization occurred after monoclonal | six weeks from monoclonal administration
  Participants will complete a questionnaire that will ask them how they felt after monoclonal antibody therapy and whether or not they required hospitalization. Medical records will be reviewed to confirm.

CONTACTS AND LOCATIONS:
Overall Officials: Sohail Rao, MD, Principal Investigator — DHR Heath Institute for Research and Development
Locations (3):
- United States (3):
  - DHR Health Institute for Research and Development, Edinburg, Texas
  - DHR Health, Edinburg, Texas
  - Starr County Memorial Hospital, Rio Grande City, Texas

IPD SHARING:
Plan to Share IPD: No